CLINICAL TRIAL: NCT06114238
Title: A Phase 1, Single-center, Open-label, Randomized, Parallel Group, Single-dose Study to Compare the Pharmacokinetics of Subcutaneous Itepekimab Administered With an Autoinjector Versus Prefilled Syringe in Healthy Participants
Brief Title: Pharmacokinetic Study to Compare Itepekimab Exposure When Administered With an Autoinjector Versus Prefilled Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKM16966; U1111-1260-3853 (Registry Identifier: ICTRP); PKM16966 (Other: Sanofi Identifier)
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — itepekimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Itepekimab administered via AI
  Interventions: Drug: Itepekimab AI
- Cohort 2 (Active Comparator): Itepekimab administered via PFS
  Interventions: Drug: Itepekimab PFS

INTERVENTIONS:
Drug: Itepekimab AI — Pharmaceutical form:Solution for injection; Route of administration: Subcutaneous AI
  Other Names: SAR440340/REGN3500
  Arms: Cohort 1
Drug: Itepekimab PFS — Pharmaceutical form:Solution for injection; Route of administration: Subcutaneous PFS
  Other Names: SAR440340/REGN3500
  Arms: Cohort 2

SUMMARY:
This Phase 1, single-center study will be conducted in an open-label, randomized, parallel design. Healthy male and female participants aged 18 to 65 years will receive a single dose of itepekimab subcutaneous (SC) administered by either a prefilled syringe (PFS) or an autoinjector (AI). Itepekimab will be administered by a trained healthcare professional (HCP).

Female and male participants will have a body weight between 50.0 and 100.0 kg and body mass index (BMI) >18.5 and ≤30 kg/m2.

Participants who satisfy the inclusion criteria will be randomized to one of the 2 study intervention groups:

* Itepekimab administered via AI (test)
* Itepekimab administered via PFS (reference) The randomization will be stratified by weight category (<70 kg, ≥70 to <80 kg and ≥80 kg) and injection site (abdomen, thigh, and arm).

Study duration for each participant is up to approximately 162 days, including:

* Screening period: up to 21 days
* Institutionalization: 2 days including 1 treatment day (Day 1)
* Follow-up period: 140 days (±5 days)
* End of study (EOS): Day 141 (± 5 days)

ELIGIBILITY:
Inclusion Criteria:

• Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

• Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameter of itepekimab: Cmax | Baseline up to EOS (approximately Day 141)
  Maximum plasma concentration of itepekimab
Assessment of PK parameter of itepekimab: AUClast | Baseline up to EOS (approximately Day 141)
  AUClast: Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast
Assessment of PK parameter of itepekimab: AUC | Baseline up to EOS (approximately Day 141)
  AUC: Area under the plasma concentration versus time curve extrapolated to infinity

SECONDARY OUTCOMES:
Assessment of PK parameter of itepekimab: tmax | Baseline up to EOS (approximately Day 141)
  Time to reach Cmax of itepekimab
Assessment of PK parameter of itepekimab: AUC0-28days | Baseline up to Day 28
  Area under the serum concentration versus time curve calculated using the trapezoidal method from time zero to 28 days
Assessment of PK parameter of itepekimab: t1/2 | Baseline up to EOS (approximately Day 141)
  Terminal half-life associated with the terminal slope (λz)
Assessment of PK parameter of itepekimab: CL/F | Baseline up to EOS (approximately Day 141)
  Apparent total body clearance of a drug from the serum
Assessment of PK parameter of itepekimab: Vss/F | Baseline up to EOS (approximately Day 141)
  Apparent Volume of Distribution at the steady state
Incidence of treatment-emergent anti-itepekimab antibodies responses | Baseline up to EOS (approximately Day 141)
Number of participants with Adverse Events (including injection site reactions), Serious Adverse Events (SAE), Adverse Event of Special Interest (AESI) | Baseline up to EOS (approximately Day 141)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Clinical Pharmacology of Miami Site Number : 8400001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM16966 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25426&tenant=MT_SNY_9011